CLINICAL TRIAL: NCT03633877
Title: A Prospective Randomized Trial of Durapore vs. Hy-Tape to Secure the Endotracheal Tube During Anesthesia.
Brief Title: Durapore vs. Hy-Tape to Secure The Endotracheal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB#: 13029
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Erythema
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Intervention Model Description: Every patient will have each tape on each side of the mouth, with Hy-Tape® on one side and DuraporeTM on the other side according to the randomization schema.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DuraporeTM on R, Hy-Tape ® on L (Experimental): DuraporeTM and Hy-Tape® will be placed on patients' skin around the mouth during general anesthesia
  Interventions: Device: DuraporeTM and Hy-Tape®
- DuraporeTM on L, Hy-Tape ® on R (Experimental): DuraporeTM and Hy-Tape® will be placed on patients' skin around the mouth during general anesthesia
  Interventions: Device: DuraporeTM and Hy-Tape®

INTERVENTIONS:
Device: DuraporeTM and Hy-Tape® — Medical tapes

SUMMARY:
While adhesive tape is commonly used to secure endotracheal tubes (ETT) during general anesthesia, its use is also associated with facial skin injuries. Although a variety of adhesive tapes are used in clinical practice, few studies have investigated the likelihood of adhesives in producing injury. The purpose of this randomized, controlled, non-inferiority study was to compare the proportion of facial skin injury with Durapore™ vs. Hy-Tape®.

DETAILED DESCRIPTION:
Adhesive tapes are often used on the patient's face during general anesthesia. They are used to fix the tracheal tube, nasopharyngeal temperature probe, nasogastric tube, and nerve stimulator electrodes. An adhesive tape used in anesthesia needs to provide fast, secure adhesion to prevent dislodgement of critical devices. The tape should be secure over time, with changes over temperature, humidity, or exposure to fluids as occurring in the operating room. However, the tape should be gentle enough that removal should not cause skin trauma to the face. While the skin irritation is generally limited to mild erythema that resolves on its own within a day or two of receiving anesthesia, the irritation may affect patient satisfaction. Furthermore, serious injury, including full-thickness epidermal loss with purpura has occurred at Tufts Medical Center with the use of 3MTM Durapore tape, requiring several doctor visits in follow up.

Medical adhesive related skin injuries are estimated to impact at least 1.5 million patients annually in the US with significant costs per incident. (1) At Tufts Medical Center, a variety of adhesive tapes are used to secure the endotracheal tube during anesthesia, including 3MTM Durapore (acrylate- based tape) and the Hy-Tape® Pink tape (zink-based tape) with no preference for one or the other.

Hy-Tape's zinc oxide-based adhesive is claimed to be soothing to delicate skin, and removes with minimum trauma, thereby reducing the chance of skin tears and tape burns. It also has the unique quality of providing maximum adhesion when it reaches body temperature, without getting more aggressive or breaking down over time as acrylic-based adhesive tapes do. However, there is no scientific evidence to support this claim.

The purpose of this study is to compare the proportion of skin erythema after general anesthesia with the use of DuraporeTM vs. Hy-Tape®.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Surgeries scheduled for anesthesia of duration more than 30 minutes after induction.

Exclusion Criteria:

1. Any patient that does not consent
2. Patients < 18 years old
3. Surgery in the prone position
4. Surgery on the head, brain, neck, teeth, mouth, eyes, or face

   Any patient who has:
5. Pre-existing skin erythema or other skin trauma
6. Lips piercings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Skin erythema | Standardized photos will be taken within 5 minutes of removing tape after surgery
  Skin photographs will be independently evaluated by three blinded dermatologists to determine presence and severity of perioral erythema. Photographs will be cropped such that only the perioral region is visible for assessment. Erythema will be evaluated on a scale of 0-3 (0 indicating none, 1 indicating mild, 2 indicating moderate, and 3 indicating severe).

SECONDARY OUTCOMES:
Skin scaling, edema, and tearing | Standardized photos will be taken within 5 minutes of removing tape after surgery
  Skin photographs will be independently evaluated by three blinded dermatologists to determine presence and severity of perioral scaling, edema, and tearing. Photographs will be cropped such that only the perioral region is visible for assessment. These outcomes will be evaluated on a scale of 0-3 (0 indicating none, 1 indicating mild, 2 indicating moderate, and 3 indicating severe).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Tsai, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No